CLINICAL TRIAL: NCT05588700
Title: A National, Multicenter, Phase III Randomized Controlled Trial to Assess the Impact of a One-year Supervised Physical Activity Program to Reduce Long-term Cancer-related Fatigue in Metastatic Testicular Germ Cell Tumor Patients
Brief Title: Impact of a Physical Activity Program to Reduce Long-term Cancer-related Fatigue in Metastatic Testicular Germ Cell Tumor Patients
Acronym: STARTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STARTER (ET 22-125)
Record Dates: First submitted 2022-10-12; First posted 2022-10-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Testicular Cancer
Keywords: fatigue; sequelae; gut microbiota composition
MeSH Terms: conditions — Testicular Neoplasms; Fatigue | interventions — Exercise; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Behavioral: Physical activity recommendations; Behavioral: Connected activity tracker
- Intervention group (Experimental)
  Interventions: Behavioral: Physical activity recommendations; Behavioral: Connected activity tracker; Behavioral: Physical Activity (PA) Intervention

INTERVENTIONS:
Behavioral: Physical activity recommendations — At the baseline, all participants will receive the international recommendations in terms of physical activity for promoting health in the general population.
Behavioral: Connected activity tracker — At baseline, all participants will receive a connected activity tracker to wear 24 hours a day during one year. Patients will be asked to download an application, dedicated to the study so that the physical activity data (ie. number of steps per day) will be synchronized in the application.
Behavioral: Physical Activity (PA) Intervention — The intervention will last 1 year and will have 2 phases. Phase 1: At each cycle of chemotherapy, patients will be proposed to perform 2-4 sessions per week. This program will be individual, supervised, performed at a moderate intensity. Between cycles, patients will be asked to perform 1-2 supervised collective live online physical activity sessions per week, proposed by a partner specialized in online PA.
  Phase 2: After chemotherapy, patients will be asked to perform 2-3 PA sessions per week at a moderate intensity. Patients will be offered 2 options of PA practice: in the supervised collective live online PA session (as already performed in the phase 1), and/or in a fitness center (this practice will take place in a "classic" environment with a 9-month free access for patients thanks to a partnership).
  In addition, patients will benefit from 4 individual motivational interviews, conducted by videoconference and/or by phone call with a professional.
  Arms: Intervention group

SUMMARY:
Testicular germ cell tumor (TGCT) is the most common malignancy in men between 15 and 40 years. Although TCGT survivors have a good survival prognosis, they suffer from short- and long-term sequelae such as chronic fatigue, psychological disorders, cardiovascular toxicities and second malignancies. The benefits of physical activity (PA) during treatments have been demonstrated in cancer patients to improve quality of life (QoL) and physical fitness and to reduce fatigue. However, few PA programs have been proposed to TGCT patients and their effects on sequelae have not been assessed yet. A growing body of evidence links treatment-related alteration in the gut microbiota to sequelae of cancer survivors, including fatigue and cardiovascular toxicities. Also, PA has been known as a possible modulator of the gut microbiota composition. To date, no study has been conducted to examine how the gut microbiota and its metabolites moderate the effect of PA on fatigue and other late effects in TGCT survivors. The objectives will be to assess the impact of a PA program on fatigue and other sequelae and to investigate how the gut microbiota and its metabolites moderate the associations between PA and sequelae. We will conduct a prospective, multicenter, phase III, randomized controlled trial of a one-year supervised PA program. 236 men with metastatic TGCT and eligible for a first line of chemotherapy will be randomly assigned to either PA intervention or control arm. All patients will benefit from a connected activity tracker and PA recommendations. In the intervention arm, PA will be based on supervised sessions and motivational interviews. The primary endpoint (fatigue) will be assessed at 3 years. The trial will provide novel insights into the impact of PA on fatigue and other sequelae in TGCT survivors with understanding a potential underlying mechanism of gut microbiota. This evidence will support the development of targeted PA guidelines to improve QoL and reduce sequelae in TGCT survivors.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years
* With a metastatic germ cell tumor histologically confirmed (seminoma and non-seminoma)
* Who have already undergone an orchidectomy
* Having a first line of chemotherapy planned with BEP, EP or VIP
* Having a smartphone (i.e. to connect the activity tracker)
* PS < or = 2
* Whose ability to practice an adapted physical activity (APA) has been certified by a medical certificate issued by the referring oncologist or the investigating physician
* Available and willing to participate in the study for the duration of the intervention and follow-up,
* Able to understand, read and write French,
* Affiliated with a social security scheme,
* Having dated and signed an informed consent.

Exclusion Criteria:

* Presence of symptomatic bone and/or brain metastases
* Central nervous system involvement with neurological deficits preventing walking
* History or coexistence of another primary cancer (apart from in situ cancer of any location and/or basal cell skin cancer and/or basal cell skin cancer and/or a cancer in complete remission for more than 3 years),
* Contraindication to physical activity (e.g. uncontrolled hypertension, uncontrolled heart disease) uncontrolled heart disease),
* Unable to be followed for medical, social, family, geographical or psychological reasons, during the entire study period,
* Deprived of liberty by judicial or administrative decision, or adults protected by law,
* Concurrent participation in another study in PA.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2031-01-14 (Estimated); Study Completion 2038-01-14 (Estimated)

PRIMARY OUTCOMES:
cancer-related fatigue, considering both physical and cognitive fatigue scores at 3 years after the start of first-line chemotherapy | Year 3
  Multidimensional aspects of fatigue will be assessed by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-FA12 cancer related fatigue module. EORTC QLQ-FA12 consists of 12 items to evaluated physical, cognitive and emotional domains of cancer-related fatigue. Participants will answer to a 4-points Likert scale ranging from "not at all" to "very much". All scores will be transformed to a 0 to 100 scale and higher scores will indicate greater degree of fatigue.
  The Primary Outcome Measure will be assessed with physical and cognitive items.

SECONDARY OUTCOMES:
other dimensions of fatigue | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  Multidimensional aspects of fatigue will be assessed by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-FA12 cancer related fatigue module. EORTC QLQ-FA12 consists of 12 items to evaluated physical, cognitive and emotional domains of cancer-related fatigue. Participants will answer to a 4-points Likert scale ranging from "not at all" to "very much". All scores will be transformed to a 0 to 100 scale and higher scores will indicate greater degree of fatigue.
  All of the secondary cancer related fatigue dimensions except the physical and cognitive items are evaluated (emotional fatigue, interference with daily life and social sequelae, assessed by the EORTC QLQ-FA12 questionnaire).
Health-related quality of life (EORTC QLQ-C30) | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  Health-Related Quality of Life (HRQoL) and fatigue will be measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ-C30). QLQ-C30 questionnaire consists of 30 items to evaluate 5 functioning domains (physical, role, emotional, cognitive, and social), a global HRQoL domain, 3 symptom domains (pain, fatigue and nausea) and 6 single items (dyspnea, insomnia, anorexia, diarrhea, constipation and financial impact).Participants will answer to a Likert scale ranging from "not at all" to "very much" and from "very bad" to "excellent" only for the global HRQoL questions. All scores will be standardized to a 0 to 100 scale according to the EORTC scoring manual. Higher scores represent better functioning, better global HRQoL and greater symptom burden.
Health-related quality of life specific for testicular cancer (EORTC QLQ-TC26) | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  The module Quality of Life Questionnaire specific to Testicular Cancer (QLQ-TC26) comprises seven multi-item scales (treatment side effects, treatment satisfaction, future perspective, communication, sexual activity, functioning and enjoyment) and six single items (job and education problems, physical limitations, family problems, infertility, body image problems, testicular transplant satisfaction).Participants will answer to a Likert scale ranging from "not at all" to "very much". All scores will be standardized to a 0 to 100 scale according to the EORTC scoring manual. Higher scores represent better functioning, better global HRQoL and greater symptom burden.
Proportion of patients who modify their cognition | Inclusion, end of chemotherapy (Month 4), Month 12, Year 2, Year 3
  The cancer-related cognitive impairment will be measured by the Functional Assessment of Cancer Therapy-Cognition (FACT-Cog). The FACT-Cog is a validated self-administrated questionnaire in order to assess memory, attention, concentration, language, and thinking abilities. The questionnaire is composed of 37 items with four subscales: patients' perceived cognitive impairments, perceived cognitive abilities, deficits observed or commented on by others, and impact of cognitive changes on HRQoL. Participant will answer how often this situation occurred during the last 7 days on a Likert-type scale ranging from "never" to "several times a day". For both scales, higher scores indicated better perceived cognitive function.
Proportion of patients who modify their anxiety and depression level | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3
  Hospital Anxiety and Depression scale (HADS) is an instrument used to screen for anxiety and depressive disorders. It has 14 rated items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score for each score = 21).
Proportion of patients who change their anthropometry | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3
  Weight (in kilograms), Height (in meters), Body Mass Index (in kg/m^2)
Physical condition and muscular strength (6-minute walk test) | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3
  assessed by the 6-minute walk test (distance traveled in meters in 6 minutes)
Physical condition and muscular strength (hand-grip) | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3
  assessed by the hand-grip test (kg)
Physical condition and muscular strength (sit-to-stand test) | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3
  assessed by the sit-to-stand test (number of repetitions)
Proportion of patients who change their physical activity (PA) and sedentary levels | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  PA and sedentary levels will be measured by National Observatory of Physical Activity and Sedentary Lifestyle - Physical Activity questionnaire (ONAPS-PAQ) This questionnaire assesses the level of physical activity and sedentary lifestyle during a typical week for the adult population. It is divided into three parts and 21 questions: activities at work, travel for utilitarian purposes and leisure or home activities. This questionnaire also assesses physical inactivity at all times of life (travel, work, leisure).
Physical activity level | Every days during the first year
  number of days wearing the tracker
Adherence to the physical activity tracker | Month 12
  number of days wearing the tracker
Satisfaction with the intervention | Month 12
  self-administered questionnaire
sleep quality and heart rate | continuously during the first year
  assessed by the connected watch
compliance with PA sessions | Month 12
  assessed by the number of sessions scheduled/performed during the different phases of the intervention
Motivation | Inclusion, end of chemotherapy (Month 4), Month 12
  This questionnaire can be used on a daily basis, for all populations, with the aim of better understanding the motivation of individuals to practice physical activities from a health perspective. The challenge is to provide professionals with an appropriate questionnaire that can assess patient motivation at the start and end of PA care.
  Participants will answer to a 7-points Likert scale ranging from "does not match at all" to "corresponds very strongly".
  This questionnaire assesses several items : intrinsic motivation, integrated regulation, identified regulation, introjected regulation, external regulation, amotivation.
  The results for each patient should be compared with the results of the validation population.
pre-intervention PA practice environment | Inclusion
  The association between the pre-intervention PA practice environment (type of activity, practice locations) and compliance with the intervention
Number of participants with neuropathies and the neuropathies level | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  Neuropathies assessed by a visual analog scale. Participants will answer to a 0 (better outcome) to 10 (worst outcome) scale.
Number of participants with pain and the pain level | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  Pain assessed by a visual analog scale. Participants will answer to a 0 (better outcome) to 10 (worst outcome) scale.
TGCT relapse | Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  CT scan/tumor-marker increase
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  Occurrence of induced-treatment toxicity according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Second primary malignancy | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  The occurence of second primary malignancy
Sustainable return to work | Month 12, Year 2, Year 3
  number of consecutive working days without sick leave
Immune and inflammatory biomarkers | Inclusion, end of chemotherapy (Month 4), Month 12, Year 3
  IL-1α/β, IL-6, IL-15, TNF-α, CRP
liver function biomarkers | Inclusion, end of chemotherapy (Month 4), Month 12, Year 3
  ALT/AST, bilirubin
gut microbiota composition and diversity | Inclusion, end of chemotherapy (Month 4), Month 12, Year 3
  measured using 16s rRNA Illumina sequencing
french validation of EORTC QLQ-TC26 | Inclusion, end of chemotherapy (Month 4), Month 6, Month 12, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  To validate the psychometric properties of the French version of the EORTC QLQ-TC26 questionnaire assessing the health-related health-related quality of life in patients with testicular cancer

CONTACTS AND LOCATIONS:
Overall Officials: Aude Fléchon, MD, Principal Investigator — Centre Leon Berard
Locations (8):
- France (8):
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - Centre Eugène Marquis, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noh H, Anota A, Mongondry R, Meyrand R, Dupuis C, Schiffler C, Marijnen P, Rinaldi S, Lachuer J, Keski-Rahkonen P, Gunter MJ, Flechon A, Fervers B, Perol O. Impact of a one-year supervised physical activity program on long-term cancer-related fatigue and mediating effects of the gut microbiota in metastatic testicular cancer patients: protocol of the prospective multicentre, randomized controlled phase-III STARTER trial. BMC Cancer. 2024 Jan 15;24(1):84. doi: 10.1186/s12885-024-11824-7. PMID 38225551